CLINICAL TRIAL: NCT02082093
Title: Medico-economic Evaluation of a Telemedicine System for the Management of Chronic Renal Failure
Acronym: eNephro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmagest Interactive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eNephro
Record Dates: First submitted 2014-02-14; First posted 2014-03-10 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; telemedicine
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Care (No Intervention)
- eNephro Application (Experimental): Telemedicine system which is a collaborative and expert system, consisting of:
  A dynamic shared medical record for the collection of administrative , medical, biological and clinical data for each patient. All health professionals can access the folder and fill in the support. It is the same for patients treated at home.
  A secure messaging for communication between health professionals and between patients and health professionals Expert systems analyzing data from each patient A management tool of therapeutic education
  These patients have a chronic renal failure moderate to end up being treated by ambulatory dialysis or kidney transplantation. The patients of each population will be randomly assigned in group 1 ie traditional care or in group 2 ie traditional care added by telemedicine system
  Interventions: Device: Telemedicine System

INTERVENTIONS:
Device: Telemedicine System
  Arms: eNephro Application

SUMMARY:
The main objective of this study is to demonstrate the efficiency ( cost-effectiveness ) of a telemedicine system : eNephro Application , compared with traditional care in the management of chronic renal failure in different populations :

* population 1 : Patients with CKD stage 3B- 4 , the combined endpoint achievement of target blood pressure and proteinuria .
* population 2 : Patients with ESRD treated by ambulatory dialysis , the cumulative duration of hospitalization in short-stay
* population 3 : Patients with ESRD treated with Renal Transplantation , the cumulative duration of unplanned short stay

Two statistical analysis will be done :

* a main analysis for the one year initial follow-up for each patient
* a secondary analysis for the one year initial follow-up estended by one year (proposed to each patient at the end of the initial follow-up), that is a 2 years period.

The intervention tested in this study is a telemedicine system which is a collaborative and expert system, consisting of:

* A dynamic shared medical record for the collection of administrative , medical, biological and clinical data for each patient. All health professionals can access the folder and fill in the support. It is the same for patients treated at home.
* A secure messaging for communication between health professionals and between patients and health professionals
* Expert systems analyzing data from each patient
* A management tool of therapeutic education

Each patient and whatever the group will perform as part of its monitoring of the CKD assessments at baseline , 6 months, 12 months, 18 months (Populations 1 and 2) and end of study (24 months). These evaluations are about compliance, quality of life, anxiety - depression state. To enhance costs the point of view retained will be health insurance's point of view. Among the various costs, only direct costs are considered: disease management, hospitalizations, consultations in hospitals and private practice, prescribed medical transportation , home visits by health professionals, additional assessments related to the evaluated intervention. A probabilistic matching with the data bases of the National Information System of the Social Insurance will be performed. In addition, the acceptability of the system of telemedicine by patients in the intervention and health professionals will be also evaluated.

DETAILED DESCRIPTION:
Three populations are recruited with the following inclusion criteria:

* age ≥ 18 years;
* ability to use a tablet device (alone or with assistance);
* population 1: stabilised stage 3B or stage 4 CKD with nephrology management of less than 3 years;
* population 2: stage 5D CKD treated by homecare peritoneal dialysis (PD) or out centre haemodialysis (HD);
* population 3: stage 5T CKD treated by renal transplantation for 3 to 12 months.

Non-inclusion criteria are:

* dialysis after renal transplantation failure;
* organ transplantation other than kidney;
* life expectancy < 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD Stage 3B 4 ESRD patients receiving ambulatory dialysis , Patients treated with Renal Transplantation
* In CKD patients stage 3B 4: nephrology care ≤ 3 years, for transplant patients: Renal Transplantation ≥ 3 months but ≤ 12 months
* Patients can use an IT tool or having in their entourage one who knows how to use

Exclusion Criteria:

* Acute Renal Failure at the time of inclusion
* Patient in transplant failure
* Patient with another organ transplant
* Patient whose life is at stake in the short term (Life expectancy <1 year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Combined endpoint achievement of target blood pressure and proteinuria | one year
  population 1 : Patients with CKD stage 3B- 4 , the combined endpoint achievement of target blood pressure and proteinuria
Cumulative duration of hospitalization in short-stay for 1 year | one year
  population 2 : Patients with ESRD treated by ambulatory dialysis , the cumulative duration of hospitalization in short-stay for 1 year
Cumulative duration of unplanned short stay for 1 year | One year
  population 3 : Patients with ESRD treated with Renal Transplantation , the cumulative duration of unplanned short stay for 1 year
Survival | One Year
  Population 2 : Survival without events event = hospitalization whatever the duration and/or return to in-center dialysis

SECONDARY OUTCOMES:
Compliance | Base Line, 6 months, One Year
  Girerd's auto questionnaire to assess compliance
Quality of Life of patients | Base Line, One Year
  Populations 1 and 2 : KDQoL questionnaire to assess quality of life Population 3 : Re TRANSQoL questionnaire
Anxiety-Depression State | Base Line, One Year
  HAD Questionnaire
Change in the glomerular filtration rate | Base Line, One Year
  Population 1 : One Year Change in the GFR estimated by MDRD equation (delta GFR/year)
Anemia Control | One Year
  the anemia control is assessed by the achievement of hemoglobin, ferritin and saturation coefficient Transferrin targets
Change in the glomerular filtration rate | Base Line, One Year
  Population 3 : One Year Change in the GFR estimated by MDRD equation (delta GFR/year)
Consultations and Hospitalizations unplanned | One Year
  Number of consultations and conventional hospitalizations unplanned in Transplantation center over a year
Disease's Costs | One Year
  To enhance cost, the health insurance's point of a view is retained. Among the various costs, only direct costs are taken into account , there are :
  * costs associated with the management of the disease
  * hospitalizations' costs
  * consultations ' costs (hospital and liberal sectors)
  * prescribed medical transport's cost
  * health professional costs
  * additional tests costs. A probabilistic matching with the data bases of the National Information System of the Social Insurance will be performed. In addition, the acceptability of the system of telemedicine by patients in the intervention and health professionals will be also evaluated.
Intervention's costs | One Year
  Costs related to the evaluated intervention : Costs installation, equipment , training and maintenance of the telemedicine system

OTHER OUTCOMES:
Acceptability | One Year
  Acceptability questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Kessler, Pr, Principal Investigator — CHU Nancy, Nephrology Service
Locations (8):
- France (8):
  - AURAD Aquitaine, Bordeaux
  - CHU Bordeaux, Bordeaux
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - TELECOM Bretagne, Brest
  - CH Dunkerque, Dunkirk
  - CHU Lille, Lille
  - ALTIR, Nancy
  - CHU Nancy, Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thilly N, Chanliau J, Frimat L, Combe C, Merville P, Chauveau P, Bataille P, Azar R, Laplaud D, Noel C, Kessler M. Cost-effectiveness of home telemonitoring in chronic kidney disease patients at different stages by a pragmatic randomized controlled trial (eNephro): rationale and study design. BMC Nephrol. 2017 Apr 5;18(1):126. doi: 10.1186/s12882-017-0529-2. PMID 28381266